CLINICAL TRIAL: NCT00078429
Title: Molecular Epidemiology of Myocardial Infarction and Stroke in Older Adults - Ancillary to CHS
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1221
Record Dates: First submitted 2004-02-25; First posted 2004-03-01 (Estimated); Last update posted 2008-07-24 (Estimated); Status verified 2008-07

CONDITIONS: Coronary Disease; Cardiovascular Diseases; Heart Diseases; Cerebrovascular Accident; Myocardial Infarction
MeSH Terms: conditions — Coronary Disease; Cardiovascular Diseases; Heart Diseases; Stroke; Myocardial Infarction

SUMMARY:
To investigation the association of thrombosis and inflammation genes with sub-clinical cardiovascular disease and with incident myocardial infarction and stroke in older adults.

DETAILED DESCRIPTION:
DESIGN NARRATIVE:

The study represents a collaborative effort among investigators of the Cardiovascular Health Research Unit, Department of Genome Sciences at the University of Washington (UW), and the multi-center Cardiovascular Health Study (CHS), including the CHS Blood Laboratory at the University of Vermont. The study links advances in thrombosis and inflammation biology, large-scale human genomics, and population and statistical genetics, with the unique resources of CHS, a large, bi-racial cohort of older adults. In older men and women without clinically apparent vascular disease, carotid intimal-medial thickness or IMT (a measure of subclinical atherosclerosis), C-reactive protein (a sensitive marker of inflammation), and D-dimer (a global marker of activation of the hemostatic system) predict subsequent clinical events such as myocardial infarction (MI) and stroke. While the therapeutic benefits of thrombolytic therapy and aspirin suggest a major role for clotting and inflammation in the etiology of coronary disease and stroke, the genetic determinants of these risk factors, which are also influenced by traditional lifestyle risk factors such as smoking and obesity, remain largely unexplored in older adults. The setting for this study is the Cardiovascular Health Study, a cohort study of 5888 older adults designed to assess risk factors for stroke and coronary disease. Data on traditional risk factors, on measures of subclinical disease, and cardiovascular events are available to the ancillary study. By integrating recent clinical and experimental data on age-related and vascular bed-specific regulation of blood coagulation, and incorporating complete human genomic DNA sequence variation data from the NHLBI-funded UW Program for Genomic Applications, the investigators will evaluate thoroughly the association of thrombosis and inflammation genes with (1) carotid IMT, CRP, and D-dimer levels measured at baseline and (2) incident MI and stroke in adults >65 years old followed for up to 12 years.

ELIGIBILITY:
No eligibility criteria

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Dates: Start 2003-07; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Reiner — University of Washington